CLINICAL TRIAL: NCT03797495
Title: Hypoplasminogenemia: An International RetroSpecTive and PrOspective CohoRt StudY (HISTORY)
Brief Title: Study of Individuals Affected With Hypoplasminogenemia
Acronym: HISTORY
Status: Recruiting | Type: Observational
Sponsor: Indiana Hemophilia &Thrombosis Center, Inc. (Other)
Collaborators: Fondazione Angelo Bianchi Bonomi (Other)
Responsible Party: Principal Investigator, Amy D Shapiro, MD, Medical Director, Indiana Hemophilia &Thrombosis Center, Inc.
Other Study IDs: HISTORY
Record Dates: First submitted 2018-12-28; First posted 2019-01-09 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2024-10

CONDITIONS: Plasminogen Deficiency
MeSH Terms: conditions — Congenital Plasminogen Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Whole blood, serum, and plasma will be retained. Time perspective is retrospective and prospective.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is an Investigator initiated retrospective and prospective single cohort study. The study will utilize an international registry and develop a specimen biobank to provide an improved understanding of the natural history of hyposplasminogenemia, to elucidate the heterogeneity of phenotypic expression, identify markers to predict disease course, and inform improved therapeutic modalities

DETAILED DESCRIPTION:
The aims of this study are to:

1. Define PLGD natural history in a large cohort of individuals with hypoplasminogenemia and their first-degree family members.
2. Identify factors that correlate with disease expression and severity.
3. Create a specimen biobank for further studies, available to other researchers.

The project will be international in scope with two collaborating centers that have created and will collect the subject data and samples. In North/Central/South America, the Indiana Hemophilia & Thrombosis Center (IHTC) will serve as the primary site while University of Milan will serve as the center for all other sites. The database is housed at the University of Milan, Italy.

Study population will include males and females affected with hyposplasminogenemia of any age. Both one-year retrospective and three-year prospective data will be collected on an international cohort of 100 affected individuals and their first degree family members (parents, siblings; total estimated study population ~500).

Study sample analysis, except for urine analyses, will be centralized and performed in Italy; the plasminogen antibody analysis will be batched for analysis, and the urine analyses will be performed locally. A sample biorepository will be created and ultimately housed in Italy. The study will provide testing for plasminogen activity and antigen, plasminogen genetic analysis, polymorphisms in genes that impact plasminogen expression and fibrinolysis, and global hemostatic assays. In addition, stored samples will be used for further testing and analyses to potentially include whole genome sequencing to further identify plasminogen genetic mutations as needed and to investigate other genetic modifiers of disease expression. An exploratory aim includes investigating the potential relationship with streptococcal strains and altered plasminogen products.

The study period will be 3 years for each enrolled subject. In-person visits will be conducted and samples for analysis will be collected at baseline and at end of study. Interval follow-up will be performed every 6 months by telephone. data will be collected at unscheduled visits that are performed for clinical need at the treating physician's discretion.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent and assent as applicable (Appendix 1)
2. A. Males or females with type 1 PD diagnosed locally with plasminogen activity levels <50% OR B. First degree family members of a person diagnosed with type 1 PD (includes parents, siblings, half-siblings)
3. All ages included
4. Available clinical history and treatment for at least 1 year prior to entry except for infants < 1 year of age
5. Willingness to provide samples for analysis including DNA, plasma etc.
6. Willingness to participate in prospective follow-up for up to 3 years

Exclusion Criteria:

1. Previous organ transplant recipient
2. Any psychiatric disorder, other mental disorder, or any other medical disorder that impairs the subject's ability to give informed consent or to comply with the requirements of the study protocol
3. Refuses to provide informed consent
4. Special patient populations, including prisoners or, are deemed medically or cognitively unsuitable for research by their treating physician
5. Inability to obtain a blood sample due to poor or limited venous access

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population will include males and females affected with hyposplasminogenemia of any age and their first degree family members (siblings and parents).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-12-18 (Actual); Primary Completion 2027-03-08 (Estimated); Study Completion 2027-04-19 (Estimated)

PRIMARY OUTCOMES:
Define the natural history of plasminogen deficiency | 2 years
  1. Recruit 100 subjects with hypoplasminogenemia and their first-degree family members
  2. Collect up to 1 year retrospective and 3 year prospective data on symptoms, treatment and interventions
Identify factors that contribute to or correlate with disease expression and severity | 5 years
  1. Perform centralized plasminogen activity and antigen analyses
  2. Perform centralized genetic analysis to identify changes in the plasminogen gene
  3. Perform centralized analysis of polymorphisms that affect plasminogen activity levels and impact fibrinolysis
  4. Perform local urine analysis
  5. Collect samples to explore the interaction of altered plasminogen proteins with bacterial strains
Create a specimen biobank | 15 years
  Bank plasma, serum and DNA on consenting enrolled subjects

CONTACTS AND LOCATIONS:
Overall Officials: Amy D Shapiro, MD, Principal Investigator — Indiana Hemophilia &Thrombosis Center, Inc.; Flora Peyvandi, MD, PhD, Principal Investigator — Univeristy of Milan
Locations (30):
- United States (12):
  - The University of Alabama (UAB), Birmingham, Alabama
  - Rush University Medical Center, Chicago, Illinois
  - Indiana Hemophila @Thrombosis Center, Indianapolis, Indiana
  - University of Minnesota, Pediatric Hem/Onc & Cancer Survivorship Program, Minneapolis, Minnesota
  - Stony Brook University | Stony Brook Medicine, East Setauket, New York
  - SUNY Upstate Medical University, Pediatric Hematology/Oncology, Syracuse, New York
  - Wake Forest University, Winston-Salem, North Carolina
  - Hemophilia Center of Western Pennsylvania, Pittsburgh, Pennsylvania
  - Vanderbilt Children's Hematology-Oncology, Nashville, Tennessee
  - Cook Children's Medical Center, Forth Worth, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Hospital Britanico Buenos Aires, Buenos Aires, Argentina
- Australia (2):
  - Murdoch Children's Research Institute, The Royal Children's Hospital, Melbourne, Victoria
  - Children's Health Queensland Hospital and Health Service, South Brisbane
- Medical University of Innsbruck, University Clinic for Pediatrics and Adolescent Medicine, Innsbruck, Austria
- Canada (4):
  - Windsor Regional Hospital, Windsor, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
  - CHU de Québec Université Laval, Québec, Quebec
  - University of Saskatchewan, Saskatoon
- Alexandra Hospital, Athens, Hematology Department, Athens, Greece
- Safra's Children Hospital, Sheba Medical Center, Tel Aviv, Israel
- Italy (2):
  - Angelo Bianchi Bonomi Hemophilia and Thrombosis Center,, Milan
  - University Hospital of Padova, Padua
- Faculty of Medicine, Chiang Mai University, Chiang Mai, Thailand
- Turkey (Türkiye) (4):
  - Dokuz Eylul University pediatric Pulmonology, Allergy and Clinical Immunology, Izmir, Balçova
  - Istanbul Üniversitesi Onkoloji Enstitüsü, Istanbul
  - Istanbul University Cerrahpsasa, Cerrahpsasa Medical Faculty Pediatric Hematology and Oncology Department, Istanbul
  - Yuzuncu Yil University Faculty of Medicine Department of Ophthalmology, Van
- Royal Free Hospital, Royal Free London NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tait RC, Walker ID, Conkie JA, Islam SI, McCall F, Mitchell R, Davidson JF. Plasminogen levels in healthy volunteers--influence of age, sex, smoking and oral contraceptives. Thromb Haemost. 1992 Nov 10;68(5):506-10. PMID 1455395
- [Background] Schuster V, Hugle B, Tefs K. Plasminogen deficiency. J Thromb Haemost. 2007 Dec;5(12):2315-22. doi: 10.1111/j.1538-7836.2007.02776.x. Epub 2007 Sep 26. PMID 17900274
- [Background] Ma Q, Ozel AB, Ramdas S, McGee B, Khoriaty R, Siemieniak D, Li HD, Guan Y, Brody LC, Mills JL, Molloy AM, Ginsburg D, Li JZ, Desch KC. Genetic variants in PLG, LPA, and SIGLEC 14 as well as smoking contribute to plasma plasminogen levels. Blood. 2014 Nov 13;124(20):3155-64. doi: 10.1182/blood-2014-03-560086. Epub 2014 Sep 10. PMID 25208887
- [Background] Celkan T. Plasminogen deficiency. J Thromb Thrombolysis. 2017 Jan;43(1):132-138. doi: 10.1007/s11239-016-1416-6. PMID 27629020
- [Background] Shapiro AD, Nakar C, Parker JM, Albert GR, Moran JE, Thibaudeau K, Thukral N, Hardesty BM, Laurin P, Sandset PM. Plasminogen replacement therapy for the treatment of children and adults with congenital plasminogen deficiency. Blood. 2018 Mar 22;131(12):1301-1310. doi: 10.1182/blood-2017-09-806729. Epub 2018 Jan 10. PMID 29321155
- [Background] Shapiro AD, Menegatti M, Palla R, Boscarino M, Roberson C, Lanzi P, Bowen J, Nakar C, Janson IA, Peyvandi F. An international registry of patients with plasminogen deficiency (HISTORY). Haematologica. 2020 Mar;105(3):554-561. doi: 10.3324/haematol.2019.241158. Epub 2020 Jan 30. PMID 32001536
- [Derived] Sang Y, Menegatti M, Brody JA, Wiggins KL, Cooley BC, Kapfer KN, Kangro K, de Laat B, Peyvandi F, Flick MJ, Smith NL, Shapiro AD, Wolberg AS. Plasminogen activation and plasmin activity are not necessary to prevent venous thrombosis/thromboembolism. Blood. 2025 Sep 11;146(11):1346-1358. doi: 10.1182/blood.2025028680. PMID 40403316